CLINICAL TRIAL: NCT06426329
Title: The Effect of Therapeutic Touch at Birth on Pain, Birth Duration, Traumatic Birth Perception and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Doç. Profesör Doktor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TR SİVAS 04
Record Dates: First submitted 2024-03-27; First posted 2024-05-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Vaginal Delivery
Keywords: Therapeutic Touch; Labor Pain; Birth Duration; Anxiety; Traumatic Birth Perception
MeSH Terms: conditions — Labor Pain; Anxiety Disorders | interventions — Therapeutic Touch; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic touch Group (Experimental): Therapeutic touch was applied twice to the women in the intervention group in addition to routine practices. The first application was performed in the latent phase of the first stage of labour, and the second was done in the active phase of labour.
  Interventions: Behavioral: Therapeutic Touch
- Standard of care Group (No Intervention): The control group did not receive any treatment.

INTERVENTIONS:
Behavioral: Therapeutic Touch — Therapeutic touch, as meaningful touch, is included in complementary medicine in the literature. It provides physical, emotional and spiritual relief, improves physiological health, makes the person feel valuable, gives confidence, peace, calmness and increases self-confidence.
  Other Names: Control Group
  Arms: Therapeutic touch Group

SUMMARY:
Aim: This study was planned to determine the effect of therapeutic touch applied at birth on pain, birth duration, traumatic birth perception and anxiety.

DETAILED DESCRIPTION:
Methods: The sample of this randomized controlled experimental research consisted of 66 (intervention group: 33; control group: 33) women. Data were collected using a Personal Information Form, Visual Analogue Scale, State Anxiety Inventory and Traumatic Childbirth Perception Scale.

ELIGIBILITY:
Inclusion Criteria:

Not having a high-risk pregnancy Having no health problems with the baby or herself Having a single foetus Being about to have a vaginal delivery Not having a chronic physical or psychiatric diagnosis Agreeing to participate in the research Not having communication and perception problems Miad (37W<) pregnancy Having with induction application

Exclusion Criteria:

having vacuum, forceps etc. intervention such as

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline
  It is a measurement tool used to evaluate pain intensity, where 0 = no pain and 10 = the most severe pain.
State Anxiety Inventory | Baseline
  It is a scale consisting of 20 items that requires the individual to answer how she feels at a certain moment and under certain conditions, taking into account her feelings about the current situation. A score of 0-19 indicates "no anxiety", 20-39 points indicates "mild", 40-59 points indicates "moderate", and 60-79 points indicates "severe anxiety".
Traumatic Birth Perception Scale | Baseline
  It consists of 13 items and measures the woman's level of perception of traumatic birth. (0-26) points: very low perception of traumatic birth (27- 52) points: low level of perception of traumatic birth (53-78) points: perception of moderately traumatic birth (79-104) points: perception of highly traumatic birth (105-130) points: very high perception of traumatic birth

SECONDARY OUTCOMES:
Visual Analogue Scale | Postpartum in 2 hour
  It is a measurement tool used to evaluate pain intensity, where 0 = no pain and 10 = the most severe pain.
State Anxiety Inventory | Postpartum in 2 hour
  It is a scale consisting of 20 items that requires the individual to answer how she feels at a certain moment and under certain conditions, taking into account her feelings about the current situation. A score of 0-19 indicates "no anxiety", 20-39 points indicates "mild", 40-59 points indicates "moderate", and 60-79 points indicates "severe anxiety".
Traumatic Birth Perception Scale | Postpartum in 2 hour
  It consists of 13 items and measures the woman's level of perception of traumatic birth. (0-26) points: very low perception of traumatic birth (27- 52) points: low level of perception of traumatic birth (53-78) points: perception of moderately traumatic birth (79-104) points: perception of highly traumatic birth (105-130) points: very high perception of traumatic birth

CONTACTS AND LOCATIONS:
Overall Officials: Sukran Ertekin Pinar, Ph.D., Principal Investigator — Cumhuriyet University
Locations (1):
- Sukran Ertekin Pinar, Sivas, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.